CLINICAL TRIAL: NCT06653296
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of ENX-102 and Determine a Dose-response for ENX-102 in Patients With Generalized Anxiety Disorder (GAD)
Brief Title: A Dose-Response Safety Study of ENX-102 in Patients With GAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENX-102-004
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: General Anxiety Disorder
Keywords: anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- ENX-102 low-dose (Experimental): ENX-102
  Interventions: Drug: ENX-102
- ENX-102 mid-dose (Experimental): ENX-102
  Interventions: Drug: ENX-102
- ENX-102 high-dose (Experimental): ENX-102
  Interventions: Drug: ENX-102

INTERVENTIONS:
Drug: ENX-102 — Four weeks of ENX-102 (0.5, 1, or 3 mg) in capsule form followed by 2 weeks of tapered dose, taken orally once daily in the evening for a 6-week total treatment period
  Other Names: ENX-102 low-dose; ENX-102 mid-dose; ENX-102 high-dose
  Arms: ENX-102 high-dose; ENX-102 low-dose; ENX-102 mid-dose
Drug: Placebo — Six weeks of placebo in capsule form taken orally once daily in the evening for a 6-week total treatment period
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of ENX-102 and determine a dose-response for the effects of ENX-102 in patients with GAD

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, inclusive of any gender identity, aged 18 to 65 years, inclusive
* Diagnosed with GAD according to the DSM-V, confirmed by MINI
* Experiencing clinically significant generalized anxiety as measured by HAM-A score ≥18 and at least moderately severe core symptoms of anxious mood and tension as measured by HAM-A Items 1 and 2, respectively, with scores each ≥2

Key Exclusion Criteria:

* Clinically predominant psychiatric diagnosis other than GAD per the MINI
* Any past/lifetime or current diagnosis of a neurocognitive disorder or psychotic disorder, or current posttraumatic stress disorder, obsessive compulsive disorder, or bipolar disorder
* Ingested prohibited medication within 5 half-lives prior to Day 1
* Current or recent moderate or severe substance use disorder as assessed by the MINI
* Unwilling or unable to abstain from alcohol or other recreational psychoactive substances such as marijuana during participation in the trial
* Has significant progressive disorders or unstable medical conditions
* Is unable to comply with the requirements of the study or, in the opinion of the Investigator, is unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks
  • Incidence and severity of treatment-emergent AEs (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Vanover, PhD, Study Director — Engrail Therapeutics INC
Locations (3):
- United Kingdom (3):
  - MAC Clinical Research, Liverpool, UK
  - MAC Clinical Research, Blackpool
  - MAC Clinical Research, Manchester

IPD SHARING:
Plan to Share IPD: No